CLINICAL TRIAL: NCT05203731
Title: The Role of Exercise in the Consolidation of Fear Extinction Learning in Adults With High Anxiety Sensitivity
Brief Title: Level of Physical Activity and Fear Learning
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 21-01657
Record Dates: First submitted 2022-01-20; First posted 2022-01-24 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-01

CONDITIONS: Generalized Anxiety Disorder; Social Anxiety Disorder; Panic Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder; Phobia, Social; Panic Disorder | interventions — Exercise; Sitting Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Participants who will be randomized to moderate intensity exercise after extinction (Day 1)
  Interventions: Behavioral: Exercise
- Seated group (Sham Comparator): Participants who will be randomized to sitting after extinction (Day 1)
  Interventions: Behavioral: Sitting

INTERVENTIONS:
Behavioral: Exercise — Moderate intensity exercise (typically a brisk walk or light run) will occur for 20 minutes after the emotional learning procedures on Day 1.
  Arms: Exercise Group
Behavioral: Sitting — Sitting will occur for 20 minutes after the emotional learning procedures on Day 1.
  Arms: Seated group

SUMMARY:
The proposed experimental study will be the first to investigate whether exercise vs. sitting enhances consolidation of extinction learning in adults with high AS and anxiety disorders, and the mechanistic pathways of expectancy, affect, and key stress response markers.

DETAILED DESCRIPTION:
This is an experimental study (not a treatment study) aiming to examine the effects of acute exercise vs. sitting on fear extinction learning in a 2-day paradigm. 50 eligible (after screening) men and women ages 18-60 with high anxiety sensitivity (AS) and an anxiety disorder (generalized anxiety disorder, panic disorder, social anxiety disorder) will participate in a consecutive 2-day paradigm. Participants will be randomized to 1 of 2 conditions immediately following the emotional learning paradigm: 1) moderate intensity exercise (n=25) or 2) sitting(n=25), for 20 minutes. Day 2 will include testing of emotional learning. Primary outcomes are physiological arousal (skin conductance, heart rate) during Day 2 procedures. Mechanistic factors, including expected negative consequences of exercise, affect during exercise, threat/shock expectancy, and changes pre-post exercise in stress related neuroendocrine markers (cortisol and alpha-amylase) and their effects on extinction recall will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 18-60
* A primary diagnosis of a DSM-5 anxiety disorder (generalized anxiety disorder, panic disorder, social anxiety disorder)
* Anxiety Sensitivity Index-3 score of ≥23 (i.e., high anxiety sensitivity)
* Able and willing to provide informed consent

Exclusion Criteria:

* Lifetime Bipolar Disorder or psychosis
* Past 3 months substance use disorder or eating disorder
* Current PTSD (past PTSD > 6 months prior to screening is allowed)
* High risk for exercise according to the Physical Activity Readiness Questionnaire and American College of Sports Medicine guidelines with excluded active medical conditions including heart conditions, lung disease, bone/joint problems, or seizures
* Women who are currently pregnant
* Acute suicide risk (active suicidal ideation with plan and intent) as indicated by a score of ≥4 on the Columbia Suicide Severity Rating Scale (C-SSRS)
* Benzodiazepine use
* Current substance abuse or positive urine toxicology screen (recreational use of marijuana is permitted based on clinical assessment on the MINI structured diagnostic interview that it does not meet criteria for cannabis use disorder)
* Stable psychiatric medications for at least 4 weeks prior to experimental procedures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Skin Conductance Response (SCR) | Day 2 Visit
  SCR will be computed for each trial by subtracting the mean skin conductance level observed during the last two seconds of context presentation from the maximal skin conductance level reached during CS presentation. All SCR values will be square-root transformed prior to any statistical analyses. To evaluate extinction recall, an extinction retention index (ERI) will be computed for each individual using the following formula: 100 - (mean SCR to the first 4 CS+E trials during recall / maximum SCR reached during conditioning for this same cue) * 100
Heart rate (HR) | Day 2 Visit
  HR will be computed for each trial by collecting Heart rate measurements during the psychophysiological procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Szuhany, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
This pilot study is not funded to support data sharing in a small pilot sample size. The Brain & Behavior Research Foundation (funder) does not require data sharing. However, individual requests for deidentified data will be considered in the future, if appropriate.